CLINICAL TRIAL: NCT00428792
Title: An Open-label, Randomized, Rater-blinded, Cross-over, Multicenter Study Comparing the Clinical Efficacy of Methylphenidate (Immediate Release/Extended Release) Treatment (20 or 40 mg Orally od) in Children With Attention-Deficit Hyperactivity Disorder (ADHD) Under Different Breakfast Conditions Over Two Weeks
Brief Title: Safety and Efficacy of Methylphenidate in Children With Attention-deficit Hyperactivity Disorder (ADHD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CRIT124DDE04
Record Dates: First submitted 2007-01-29; First posted 2007-01-30 (Estimated); Results first posted 2011-05-06 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-04

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: ADHD; methylphenidate; children; food effect; Attention-Deficit Hyperactivity Disorder (ADHD) in children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Very light breakfast (VLB) then standard breakfast (SB) (Experimental): Very light breakfast (VLB) for one week then crossover to standard breakfast (SB) for one week while taking either 1 or 2 20 mg capsules of methylphenidate once per day based on the dosage the child had taken in the month prior to study start. VLB is defined as 150 kcal for children age 6-9 and 180 kcal for children age 10-12. SB is defined as 450 kcal for girls age 6-9, 490 kcal for boys age 6-9, 550 kcal for girls age 10-12, and 600 kcal for boys age 10-12.
  Interventions: Drug: Methylphenidate 20 mg long-acting capsules
- Standard breakfast (SB) then very light breakfast (VLB) (Experimental): Standard breakfast (SB) for one week then crossover to very light breakfast (VLB) for one week while taking either 1 or 2 20 mg capsules of methylphenidate once per day based on the dosage the child had taken in the month prior to study start. SB is defined as 450 kcal for girls age 6-9, 490 kcal for boys age 6-9, 550 kcal for girls age 10-12, and 600 kcal for boys age 10-12. VLB is defined as 150 kcal for children age 6-9 and 180 kcal for children age 10-12.
  Interventions: Drug: Methylphenidate 20 mg long-acting capsules

INTERVENTIONS:
Drug: Methylphenidate 20 mg long-acting capsules
  Other Names: Ritalin LA

SUMMARY:
This study evaluated the safety and clinical effect of treatment with methylphenidate under different breakfast conditions (minimal breakfast versus standard continental breakfast) in children with Attention-Deficit Hyperactivity Disorder (ADHD).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-12
* Diagnosis of Attention-Deficit Hyperactivity Disorder (ADHD)
* Current medication with either 20 mg or 40 mg immediate release methylphenidate

Exclusion Criteria:

* Concomitant psychiatric disorders requiring pharmacological treatment
* Concomitant severe somatic disorders
* Eating disorders
* Addiction disorders
* Very high or low body weight according to age
* Known hypersensitivity to methylphenidate
* Contraindications for methylphenidate

Other protocol-defined inclusion/exclusion criteria applied to the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2007-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharma, Study Chair — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Freiburg im Breisgau, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Very Light Breakfast (VLB) Then Standard Breakfast (SB): Very light breakfast (VLB) for one week then crossover to standard breakfast (SB) for one week while taking either 20 mg or 40 mg capsules of methylphenidate once daily based on the dosage the child had taken in the month prior to study start. VLB is defined as 150 kcal for children age 6-9 and 180 kcal for children age 10-12. SB is defined as 450 kcal for girls age 6-9, 490 kcal for boys age 6-9, 550 kcal for girls age 10-12, and 600 kcal for boys age 10-12.
- Standard Breakfast (SB) Then Very Light Breakfast (VLB): Standard breakfast (SB) for one week then crossover to very light breakfast (VLB) for one week while taking either 20 mg or 40 mg capsules of methylphenidate once daily based on the dosage the child had taken in the month prior to study start. SB is defined as 450 kcal for girls age 6-9, 490 kcal for boys age 6-9, 550 kcal for girls age 10-12, and 600 kcal for boys age 10-12. VLB is defined as 150 kcal for children age 6-9 and 180 kcal for children age 10-12.
Period: Overall Study
Arm/Group | Very Light Breakfast (VLB) Then Standard Breakfast (SB) | Standard Breakfast (SB) Then Very Light Breakfast (VLB)
Started | 80 | 70
Completed | 79 (Information is not available during which cross-over period patients discontinued.) | 66 (Information is not available during which cross-over period patients discontinued.)
Not Completed | 1 | 4
Not completed — Lack of Efficacy | 1 | 3
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Very Light Breakfast (VLB) Then Standard Breakfast (SB) | Standard Breakfast (SB) Then Very Light Breakfast (VLB) | Total
Number analyzed (Participants) | 80 | 70 | 150
Age Continuous [Mean (Standard Deviation); unit: years] — Safety Population
  years | 9.6 (1.6) | 9.7 (1.5) | 9.7 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Population
  Participants
    Female | 25 | 13 | 38
    Male | 55 | 57 | 112

OUTCOME MEASURES:

1. Primary Outcome: Fremdbeurteilungsbogen für Aufmerksamkeitsdefizit-Hyperaktivitätsstörungen (FBB-AHDS) Teacher Rating in the Intent-to-Treat (ITT) Population
Description: The FBB-ADHS is a 20-item rating scale. Each item describes a typical ADHD symptom. The 20 items are divided into 3 subscales: Attention deficits (9 items), hyperactivity (7 items), and impulsiveness (4 items). Each item is rated on a scale of 0 = not at all up to 3 = very much. The FBB-ADHS was completed by teachers on Friday afternoon of each week of the study. A total score (sum of all items divided by 20) was calculated. The total score can range from 0 to 3. A lower score indicates more ADHD.
Time Frame: Friday of each of the 2 treatment weeks
Population: Intent to treat (ITT) population: All randomized patients with at least one post-baseline measurement of the primary endpoint in both study periods.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Very Light Breakfast (VLB) Treatment Group: Very Light Breakfast (VLB) for one week while taking either 20 mg or 40 mg capsules of methylphenidate once daily based on the dosage the child had taken in the month prior to study start. VLB is defined as 150 kcal for children age 6-9 and 180 kcal for children age 10-12. SB is defined as 450 kcal for girls age 6-9, 490 kcal for boys age 6-9, 550 kcal for girls age 10-12, and 600 kcal for boys age 10-12.
- Standard Breakfast (SB) Treatment Group: Standard breakfast (SB) for one week while taking either 20 mg or 40 mg capsules of methylphenidate once daily based on the dosage the child had taken in the month prior to study start. SB is defined as 450 kcal for girls age 6-9, 490 kcal for boys age 6-9, 550 kcal for girls age 10-12, and 600 kcal for boys age 10-12. VLB is defined as 150 kcal for children age 6-9 and 180 kcal for children age 10-12.
Arm/Group | Very Light Breakfast (VLB) Treatment Group | Standard Breakfast (SB) Treatment Group
Number analyzed (Participants) | 144 | 144
Units on a scale | 0.97 (0.63) | 1.01 (0.63)

2. Secondary Outcome: Fremdbeurteilungsbogen für Aufmerksamkeitsdefizit-Hyperaktivitätsstörungen (FBB-AHDS) Attention Deficit Subscale Teacher Rating
Description: Teacher rating of the attention deficit subscale (9 items), one of 3 subscales in the FBB-ADHS. Each item is rated on a scale of 0 = not at all up to 3 = very much. The rating was completed by teachers on Friday afternoon of each week of the study. A total score (sum of all items divided by 9) was calculated. The total score can range from 0 to 3. A lower score indicates more ADHD.
Time Frame: Friday of each of the 2 treatment weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Very Light Breakfast (VLB) Treatment Group | Standard Breakfast (SB) Treatment Group
Number analyzed (Participants) | 144 | 144
Units on a scale | 1.19 (0.68) | 1.23 (0.69)

3. Secondary Outcome: Fremdbeurteilungsbogen für Aufmerksamkeitsdefizit-Hyperaktivitätsstörungen (FBB-AHDS) Hyperactivity Subscale Teacher Rating
Description: Teacher rating of the hyperactivity subscale (7 items), one of 3 subscales in the FBB-ADHS. Each item is rated on a scale of 0 = not at all up to 3 = very much. The rating was completed by teachers on Friday afternoon of each week of the study. A total score (sum of all items divided by 7) was calculated. The total score can range from 0 to 3. A lower score indicates more ADHD.
Time Frame: Friday of each of the 2 treatment weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Very Light Breakfast (VLB) Treatment Group | Standard Breakfast (SB) Treatment Group
Number analyzed (Participants) | 144 | 144
Units on a scale | 0.72 (0.70) | 0.75 (0.69)

4. Secondary Outcome: Fremdbeurteilungsbogen für Aufmerksamkeitsdefizit-Hyperaktivitätsstörungen (FBB-AHDS) Impulsiveness Subscale Teacher Rating
Description: Teacher rating of the hyperactivity subscale (4 items), one of 3 subscales in the FBB-ADHS. Each item is rated on a scale of 0 = not at all up to 3 = very much. The rating was completed by teachers on Friday afternoon of each week of the study. A total score (sum of all items divided by 4) was calculated. The total score can range from 0 to 3. A lower score indicates more ADHD.
Time Frame: Friday of each of the 2 treatment weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Very Light Breakfast (VLB) Treatment Group | Standard Breakfast (SB) Treatment Group
Number analyzed (Participants) | 144 | 144
Units on a scale | 0.93 (0.92) | 0.99 (0.90)

5. Secondary Outcome: Fremdbeurteilungsbogen für Aufmerksamkeitsdefizit-Hyperaktivitätsstörungen (FBB-AHDS) Parent Rating
Description: as for outcome 1
Time Frame: Saturday of each of the 2 treatment weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Very Light Breakfast (VLB) Treatment Group | Standard Breakfast (SB) Treatment Group
Number analyzed (Participants) | 143 | 144
Units on a scale | 1.15 (0.60) | 1.11 (0.55)

6. Primary Outcome: Fremdbeurteilungsbogen für Aufmerksamkeitsdefizit-Hyperaktivitätsstörungen (FBB-AHDS) Teacher Rating in the Per Protocol (PP) Population
Description: as for outcome 1
Time Frame: Friday of each of the 2 treatment weeks
Population: Per protocol (PP) population: All patients in the ITT population who (a) met the inclusion/exclusion criteria liable to affect the efficacy assessment and (b) did not violate the protocol in a manner liable to affect the efficacy assessment.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Very Light Breakfast (VLB) Treatment Group | Standard Breakfast (SB) Treatment Group
Number analyzed (Participants) | 131 | 131
Units on a scale | 0.93 (0.62) | 1.0 (0.63)

7. Secondary Outcome: 10-Minute Math Test - Problems Attempted
Description: The 10-Minute Math Test is a paper and pencil test consisting of several pages of math problems requiring addition, subtraction, multiplication and division calculations presented in ascending order of difficulty during a 10-minute period. Test difficulty was altered for subjects at different skill levels and ages. The number of problems attempted is an objective measure related to "academic productivity". The math test was carried out on the Saturday visit at the end of each of the 2 treatment weeks under supervision of a teacher who had been trained on this test.
Time Frame: Saturday of each of the 2 treatment weeks
Population: Intent to treat (ITT) population includes all randomized patients with at least one post-baseline measurement of the primary endpoint in both study periods. Following the intent-to-treat principle, patients were analyzed according to the treatment they were assigned to at randomization.
Measure: Mean (Standard Deviation); unit: Problems attempted
Arm/Group | Very Light Breakfast (VLB) Treatment Group | Standard Breakfast (SB) Treatment Group
Number analyzed (Participants) | 142 | 142
Problems attempted | 116.3 (56.14) | 118.1 (57.74)

8. Secondary Outcome: 10-Minute Math Test - Problems Solved
Description: as for outcome 7
Time Frame: Saturday of each of the 2 treatment weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Problems solved
Arm/Group | Very Light Breakfast (VLB) Treatment Group | Standard Breakfast (SB) Treatment Group
Number analyzed (Participants) | 142 | 142
Problems solved | 106.7 (58.34) | 108.6 (60.67)

9. Secondary Outcome: Clinical Global Impression Severity (CGI-S) Scale Score - Physician Rating of Severity
Description: The CGI-S is a scale to assess the global severity of illness. The rating is determined by the investigator answering one question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" Ratings are on a 7-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients. The rating is based upon the average observed and reported symptoms, behavior, and function in the past 7 days.
Time Frame: Saturday of each of the 2 treatment weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Very Light Breakfast (VLB) Treatment Group | Standard Breakfast (SB) Treatment Group
Number analyzed (Participants) | 142 | 143
Units on a scale | 2.75 (1.45) | 2.74 (1.48)

10. Secondary Outcome: Clinical Global Impression (CGI-I) Scale Score - Physician Rating of Improvement (Change in State)
Description: The CGI-I is a scale to assess improvement (change in state) of illness. The rating is based on the investigator answering one question: "Compared to the patient's condition prior to medication, this patient's condition is: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment." The investigator compares the patient's overall clinical condition to the 1 week period just prior to the initiation of medication.
Time Frame: Saturday of each of the 2 treatment weeks
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Very Light Breakfast (VLB) Treatment Group | Standard Breakfast (SB) Treatment Group
Number analyzed (Participants) | 142 | 142
Units on a scale | 3.49 (1.08) | 3.56 (1.18)

ADVERSE EVENTS:
Description: Safety population: All randomized patients who took at least 1 dose of study drug in 1 of the 2 treatment periods.
Arm/Group | Very Light Breakfast (VLB) Then Standard Breakfast (SB) | Standard Breakfast (SB) Then Very Light Breakfast (VLB)
Serious Adverse Events (participants affected / at risk) | 0/148 | 0/149
Other Adverse Events (participants affected / at risk) | 0/148 | 0/149

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.